CLINICAL TRIAL: NCT05235477
Title: Clinical Evaluation of the Use of Surgical Tube Technique Versus Hyaluronic Acid Gel Injection in Reconstruction of the Interproximal Papilla in Patients With Class II Papillary Deficiency
Brief Title: Clinical Evaluation of the Use of Surgical Tube Technique Versus Hyaluronic AcidInjection in Reconstruction of the Interproximal Papilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: waleed mohammad sabry (Other)
Responsible Party: Sponsor-Investigator, waleed mohammad sabry, lecturer Assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11621
Record Dates: First submitted 2022-01-03; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: the Clinical Effect of Surgical Tube Technique in Reconstruction of the Interproximal Papilla
MeSH Terms: interventions — Cell Migration Assays, Leukocyte

STUDY DESIGN:
Intervention Model Description: Group A (Intervention): Patients will receive Tube technique. Group B (Control): Patients will receive Hyaluronic acid.
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention only the outcome assessor and the statistician will be blinded.
  Single blinded:
  * Blinding of the participants is not applicable.
  * Blinding of the operator is not applicable.
  * Outcome assessor (primary and secondary outcomes) and biostatistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tube technique. (Experimental): The excavator is used to do the same on the palatal aspect. The recipient site at this time should resemble a "tube" with two openings; one on the buccal aspect at the mucogingival junction and one on the palatal aspect. To harvest the graft, the incision is made parallel to and 2 mm away from the gingival margin. A thin flap containing the keratinized tissue is separated, then the second incision is made parallel to the gingival margin, but perpendicular to the alveolar bone. With a sharp periosteal elevator, the graft is raised with the periosteum and released at its anterior and posterior ends, and then from its base .
  Interventions: Procedure: Tube technique
- Hyaluronic acid. (Active Comparator): The product used in this trial is Restylane Lidocaine (Restylane-Lidocaine cross-linked Hyaluronic Acid Filler, Galderma S.A, Sweden). Restylane was the first FDA-approved HA filler in 2003. Restylane is a non-animal stabilised cross-linked HA filler with an HA concentration of 20 mg/ml. It is a minimally invasive non-surgical injection of hyaluronic acid that observed to overcome the major limiting factor in most surgical techniques regarding the limited blood supply and the small working space. Supported by a recent study conducted by Jinng etal. 2019, who reported significant increase in the height of the gingival papilla and reduction of the area of the black triangle between baseline and 3 or 6 months in a group with thick gingival biotype after injection with hyaluronic acid, that was adding possible maximum effect with minimal postoperative hazards.
  Interventions: Procedure: Tube technique

INTERVENTIONS:
Procedure: Tube technique — An excavator (smaller than the width of the defect; evaluated pre-surgically on a study model) is used to carefully reflect the papilla away from the alveolar bone and root surfaces on the buccal aspect to access the interproximal region to prepare the bed for the graft. The excavator is used to do the same on the palatal aspect. The amount of reflection should yield a very relaxed papilla flap that permits placement of the papilla at the new coronal position without tension. The recipient site at this time should resemble a "tube" with two openings; one on the buccal aspect at the mucogingival junction and one on the palatal aspect.

SUMMARY:
Restoring defective interdental papilla partially or totally in structure and function creates a challenge in dental field owing to the small working space and limited blood supply to the area.

This led to the innovation of different techniques for treatment of defective interdental papilla that aimed at papillary tissue augmentation reported to be attained through influencing connective tissue cell proliferation, providing clot stability, protecting the reconstructed site during wound healing.

Among these techniques is the injection of hyaluronic acid gel have been considered of the latest non-invasive technique to escape drawbacks of surgeries. Though proved to have some positive results in the literature however still entails unpredicted complete gingival papilla improvement because of the diverse injection methods, cycles, dosage, and the course of treatment that needs further optimization, in addition to the lack of unified patient inclusion criteria, especially the gingival biotype .

Several surgical techniques designed to host the richest effective known sub-epithelial connective tissue graft had failed to allow maximum benefit of the graft due to the disadvantages from the number and location of incisions of their flap design, which possibly disrupt the blood supply needed added to unconsidered flap thickness, and flap retraction that impacted the success of soft tissue grafting.

Surgical Tube technique has recently been developed optimizing flap thickness, flap retraction and tension to escape disturbance of the blood supply of the graft by its use of apical incisions and containment of the graft within a rich vascular enclosed bed, thereby offering an attempt to guarantee integrity of soft tissue with no disruption of blood supply.

DETAILED DESCRIPTION:
The interdental papilla is the gingival portion that fills the proximal area under the contact between two adjacent teeth, where it is defined as gingival tissues extending from incisal tip of the papilla to a line tangential to the adjacent margins of the adjacent teeth. Anatomically, it is small and delicate with a diminutive blood supply, it is almost the most important esthetic part during smiling.

Nordland & Tarnow 1998 classified papillary loss according to system which utilizes 3 identifiable anatomical landmarks: the interdental contact point, the facial apical extent of the cemento-enamel junction (CEJ) and the interproximal coronal extent of the CEJ. Normal Interdental papilla fills embrasure space to the apical extent of the interdental contact point/area. Class I which the tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the interproximal CEJ (space present but interproximal CEJ is not visible). Class II which the tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial CEJ (interproximal CEJ visible). Class III which the tip of the interdental papilla lies level with or apical to the facial CEJ.

The absence of interdental papilla contributes to chronic retention of food debris leading to subsequent affection of periodontal health and esthetically unaccepted black triangle. To be influenced by the initial position of the teeth (diastema), the length of gingival niche area, triangular shaped crown, divergent roots and periodontal bone loss. Also tooth brush trauma and decreased keratinization due to ageing has also been implicated as a causative factor of interdental papilla loss.

Reconstruction of papillary insufficiency is one of the most difficult and challenging periodontal treatments. This is because the interdental papilla is a small, fragile area with minor blood supply which seems to be the major limiting factor in all surgical and augmentation techniques.

The injection of biocompatible hyaluronic acid gel (HA) have been considered conventional non-invasive techniques for treatment of deficient papilla. Hyaluronic acid (0.1) mm It is an essential glycosaminoglycan of the extracellular matrix of the periodontal tissues, and the majority of cells can produce it during several phases of their cell cycle. It is involved in tissue repair and wound healing by stimulating cell proliferation, migration and interaction with several growth factors. Furthermore, HA has a crucial role in space-filling owing to its hygroscopic nature. Moreover, it regulates osmotic pressure and enhances tissue lubrication and resiliency, which helps in maintaining the structural and homeostatic integrity of tissues.

However, hyaluronic acid gel injection still entails unpredicted complete gingival papilla improvement owing to the relative compact nature of the gingiva and influence of the gingival biotype that could hinder the positive outcomes on favor of thick biotype that could help to enrich the effect of hyaluronic acid through accelerating the thick connective tissue related abundance of gingival fibroblast proliferation, promoting the generation of collagen fibers. Limited studies have utilized HA gels for papillary reconstruction but still lacking a high degree of evidence and predictability.

Several conventional surgical approaches using traditional periodontal plastic and augmentation procedures aiming for complete papilla fill to overcome this problem. However, flap design were found to be invasive with increased patient morbidity, limited success, long-term stability and unpredictability due to small working spaces and limited blood supply.

Most of the surgical approaches targeting papilla reconstruction were based on Sub-epithelial connective tissue graft. Han & Takei 1996 used semilunar coronally repositioned papilla based on the use of free connective tissue graft. He concluded that subsequent second- and possibly third-stage surgery should reconstruct more of the papilla which is considered one of the disadvantages of this flap design. So Pellegrine 1996 modified this technique by folding the CTG to provide adequate thickness of the attached gingiva.

Modified Beagle's technique and Beagle's surgical technique were unpredictable due to small working spaces and limited blood supply to the area in addition to the vertical releasing incisions that could further jeopardize vascular supply and leave unpleasant scarring after healing.

Han and Tackei technique made a trial to modify the flap design by semilunar coronally repositioned papilla that enabled to preserve the interdental papilla blood supply and improving the gingival biotype from 0.75 mm to 2 mm, One year post-operative view showing 80% papillary fill.

These subepithelial conventional techniques were unpredictable due to small working spaces and limited blood supply to the area. Disadvantages of these techniques were mostly due to the number and location of incisions, which could have disrupted the blood supply needed for complete healing.

Microsurgical techniques had been introduced and enhance the visual accuracy by means of illumination and magnification. Literature on periodontal microsurgery showed improved surgical outcome when used for root coverage procedure and regenerative therapy. By the aid of subepithelial connective tissue, the microsurgical technique found to maintain the reconstructed papilla remained stable and without any clinical signs of inflammation for 4 years after surgical procedure, but the long-term survivability and the technique sensitivity involved in the surgery are to be considered.

Recent clinical study assessed the efficacy of microsurgical reconstruction of lost interdental papillam and was based on single surgical intervention, with the aid of connective tissue graft which is proved useful in Correction of papillary loss, but the Maximum gain with single procedure was found to be limited. Other limitations of the study were being due to smaller sample size and short period of follow up and were recorded for long term clinical and histological follow up studies are necessary before its predictability.

Tube technique is recently introduced by Hooshang etal. 2020 on the track of surgical techniques to overcome disadvantages of the other techniques. The innovated flap design of tube technique does not disturb the blood supply of the graft by its use of apical incisions and containment of the graft within a rich vascular enclosed bed, thereby offering reliable and satisfactory results. Integrity of the soft tissue is key to the successful outcome of this technique. The tube grafting technique requires technical precision. It is sensitive to any surgical trauma and tension, especially when the recipient site tissue is delicate.

Thus, the present randomized clinical trial is to compare the clinical effect of surgical Tube technique versus Hyaluronic Acid Gel injection in Reconstruction of the interproximal papilla in patients with class II papillary defect.

ELIGIBILITY:
Inclusion Criteria:

* Highly motivated patients with papillary deficiency types II, according to Nordland and Tarnow 1998 classification will be selected, having at least one deficient papilla in the anterior region.

  * Distance between the contact point and inter-proximal bone crest (CP-BC) of ≤ 7 mm and probing depth of ≤ 4 mm at the deficient papillary site (Abdelraouf etal. 2019).
  * Patients with full mouth plaque index (PI) and gingival index (GI) scores should be between 0-1.
  * Healthy patients free of any medical condition.

Exclusion Criteria:

* ● Patients with medical conditions that may affect periodontal healing or regeneration.

  * Patients with a history of allergic reactions, pregnant or breastfeeding females, smokers and alcoholics.
  * Patients with current or previous drugs intake that may predispose to gingival enlargement.
  * Patients under orthodontic treatment or had orthodontic treatment in the past six months.
  * Carious teeth, proximal restorations or fixed prosthesis.
  * Patients with a history of traumatic oral hygiene measures or periodontal surgeries over the last six months at the area of interest or having any scar tissue.
  * Poor oral hygiene patients.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
interdental papilla loss (Decrease of black triangle area ) (mm2) | 6 months
  The surface area of the black triangle (SABT) is assessed using standardized digital clinical photographs analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA). The surface area of the black triangle was assessed from the photographs taken at baseline (before injection), 3 and 6 months from the first injection.
  - 10 mm William's graduated periodontal probe was used as a scale for calibration.

SECONDARY OUTCOMES:
Gain in papillary height | 6 months
  Papilla Presence Index (PPI) by periodontal probe

OTHER OUTCOMES:
CAL | 6 months
  CAL will be determined by measuring the distance from the cemento-enamel junction to the base of the pocket using a UNC 15 periodontal probe.
PD | 6 months
  Probing depth will be measured from the gingival margin to the base of the periodontal pocket using a UNC 15 periodontal probe
GR | 6 month
  Gingival recession will be measured using UNC periodontal probe from the cemento-enamel junction till the gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- Waleed Mohammad Sabry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-06-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT05235477/Prot_000.pdf